CLINICAL TRIAL: NCT06662266
Title: Prospective Evaluation of Induce XT™ Bone Graft in Foot and Ankle Fusion
Brief Title: Induce XT™ Bone Graft in Foot and Ankle Fusion
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Red Rock Regeneration Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-NMP-005
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Surgery; Foot Deformities; Ankle Arthropathy
MeSH Terms: conditions — Foot Deformities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diverse group of participants who require hindfoot or ankle arthrodesis (Other): The selection criteria are designed to ensure that the study population represents the typical patients undergoing these procedures.
  Interventions: Device: Induce XT™ is a mixture of human cortical bone fibers and microparticulates that have been processed into Natural Matrix Protein® (NMP®) to which cancellous bone microparticulates have been added

INTERVENTIONS:
Device: Induce XT™ is a mixture of human cortical bone fibers and microparticulates that have been processed into Natural Matrix Protein® (NMP®) to which cancellous bone microparticulates have been added — Bone graft material is required for successful foot and ankle fusion surgery. Current bone grafting materials include autogenous bone, Augment Bone Graft and demineralized bone matrix (DBM), each of which have limitations.
  Induce XT is a novel bone graft material that can potentially be used in foot and ankle fusions that may overcome some of these limitations.

SUMMARY:
The goal of this study is to evaluate how effective Induce XT is in patients undergoing foot and/or ankle surgery. Induce XT is a bone graft material used in surgeries to fill gaps where bone is missing, such as during foot and ankle fusion. Participants in the study will have a screening visit to determine eligibility, followed by an assessment on the day of surgery and 5 follow-up visits over 12 months. These visits will include X-rays, pain evaluations, and questionnaires.

DETAILED DESCRIPTION:
Clinical Background Ankle and hindfoot arthrodesis (fusion) is a well-established treatment for various foot and ankle conditions. These surgeries require supplemental graft material. Autogenous bone graft (ABG), typically harvested from sites like the iliac crest bone graft (ICBG), is considered the gold standard for bone grafting. However, the use of ABG presents several challenges, such as increased surgical time, blood loss, and the risk of infection and pain at the donor site. Additionally, the supply of autogenous bone is limited (Boone 2003, Baumhauer, Glazebrook et al. 2020).

Augment® Bone Graft is a substitute used to enhance bone healing in foot and ankle surgeries. It contains recombinant human platelet-derived growth factor BB (rhPDGF-BB) and a beta-tricalcium phosphate (β-TCP) matrix. The β-TCP matrix provides a structure that supports new bone growth, while rhPDGF-BB stimulates the recruitment and proliferation of cells involved in bone formation and promotes both angiogenesis and bone healing. Studies have demonstrated that Augment Bone Graft can be an alternative to ABG in foot and ankle fusion procedures (DiGiovanni, Lin et al. 2013). However, Augment is costly, must be stored at 2 to 8°C, and may handle poorly. It should also not be used in patients with cancer, near resected tumors, or in those who are pregnant or may become pregnant. Additionally, the radiopaque nature of β-TCP can obscure radiographic images, making it difficult to assess bone healing (FDA 2015, FDA 2018).

Demineralized bone matrix (DBM) is another option, used alone or in combination with ABG to support bone fusion. DBM provides a scaffold for new bone growth (osteoconduction) and has osteoinductive properties due to the presence of bone morphogenetic proteins (BMPs), including BMP-2. DBM also contains growth factors that promote angiogenesis and bone formation. However, its clinical effectiveness is limited due to the low amount and bioavailability of growth factors (Gruskin, Doll et al. 2012).

Study Rationale Induce XT is a new bone matrix product combining Natural Matrix Protein® (NMP®) derived from demineralized human cortical bone allograft with mineralized cancellous bone allograft. NMP has demonstrated higher bioavailability of BMP-2 and BMP-7 and enhanced osteoinductive activity compared to DBM in various studies (Kohen, Shivanna, and Peel 2022, Peel 2023). The mineralized cancellous bone component provides additional compression resistance and allows the graft to be seen on radiographs immediately after implantation. Induce XT is clinically used as a bone void filler.

Since its market release in January 2022, NMP bone grafts have been used in over 7,500 surgeries, including spine and foot/ankle fusions, with no reported adverse events. A retrospective study also showed a high fusion rate in lumbar spine procedures using NMP fibers (Nunley 2024).

This prospective clinical trial will enroll 60 patients at one clinical site in Canada to evaluate the safety and efficacy of Induce XT in hindfoot or ankle fusion surgeries. The study will assess radiographic, clinical, functional, and quality-of-life outcomes over a 52-week postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting all of the following criteria will be considered eligible for study participation:

  1. Patient has a bone defect in the hindfoot or ankle; and
  2. Is requiring fusion using an open surgical technique with supplemental bone graft/substitute; and
  3. Fusion site is able to be rigidly stabilized with no more than 3 screws across the fusion site; and
  4. Patient is requiring one of the following procedures:

     * Ankle joint fusion
     * Subtalar fusion
     * Calcaneocuboid fusion
     * Talonavicular fusion
     * Triple arthrodesis (subtalar, talonavicular and calcaneocuboid joints)
     * Double fusions (talonavicular and calcaneocuboid joints).

Exclusion Criteria:

* Patient meeting any of the following criteria will be excluded from study participation:

  1. Patient is under 18 years of age at the time of consent;
  2. Patient has an active (local or systemic) infection or is undergoing adjunctive treatment for infection;
  3. Patient has previous fusion surgery of the proposed fusion site;
  4. Patient has cognitive disorders or is unable to complete questionnaires or provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Bone Fusion | At 24 and 52 weeks
  Fusion as measured by X-Ray
Percent bridging bone | At 24 and 52 weeks
  Measured by Computerized Tomography (CT)

SECONDARY OUTCOMES:
Disability score for foot and ankle condition | At 24 and 52 weeks
  Measured by American Orthopedic Foot and Ankle Society (AOFAS) score 0 to 100 with higher score showing better outcome
Patient reported health survey | At 24 and 52 weeks
  Measured by The Veterans RAND 12-Item Health Survey (VR-12) questionnaire- a self-reported assessment of health with higher scores indicating better perceived health

OTHER OUTCOMES:
Pain upon weight bearing | At 24 and 52 weeks
  Measured by Visual Analogue Scale (VAS) measured from 0 to 100 with lower score
Pain at fusion site | At 24 and 52 weeks
  Measured by Visual Analogue Scale (VAS) measured from 0 to 100 with lower score indicating less pain
Device related Serious Adverse Events | Day of Surgery up to 52 weeks
  Measured by clinical assessment and patient reported symptoms
Incidence of re-operation | Day of Surgery up to 52 weeks
  Secondary surgical intervention undertaken to promote fusion

CONTACTS AND LOCATIONS:
Overall Officials: Sean Peel, Study Director — Red Rock Regeneration Inc.
Locations (1):
- Halifax Infirmary, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No